CLINICAL TRIAL: NCT04966962
Title: Establishment and Validation of an Early Diagnostic Model for Bladder Cancer Based on Serum and Urine Metabolomics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); The Seventh Affiliated Hospital of Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SysMU-diag1
Record Dates: First submitted 2021-07-09; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; metabolomics
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bladder cancer: Patients who diagnosis with incident or recurrent bladder cancer
  Interventions: Diagnostic Test: serum and urine metabolomics
- benign disease of urinary system: Patients who clinically diagnosis with benign disease of the urinary system, such as urinary calculi and benign prostatic hyperplasia.
  Interventions: Diagnostic Test: serum and urine metabolomics

INTERVENTIONS:
Diagnostic Test: serum and urine metabolomics — serum and urine samples will be collected for metabolomics analysis

SUMMARY:
Metabolomics is a complementary approach for identifying perturbed metabolic pathways. The goal of this study is to establish and validate an early diagnostic model for bladder cancer by metabolomics.

DETAILED DESCRIPTION:
Early diagnosis and life-long surveillance are clinically important to improve the long-term survival of bladder cancer patients. Currently, a noninvasive biomarker that is as sensitive and specific as cystoscopy in detecting bladder cancer is lacking. Metabolomics are small organic molecules (below 2000 mass units) that are products of complex pathways. This is a prospective study aims to create an early diagnostic model based on serum and urine metabolomics. Commonly employed metabolomics analytical platforms include nuclear magnetic resonance spectroscopy (NMR), gas chromatography mass spectrometry (GC-MS), and liquid chromatography mass spectrometry （LC-MS）. The diagnostic model will be made to distinguish bladder cancer and benign disease of the urinary system.

ELIGIBILITY:
Inclusion Criteria:

Bladder cancer group:

1. Any male or female patient aged 18 or older
2. Able to provide serum and urine specimen before treatment
3. Diagnosis with incident or recurrent bladder cancer

Control group

1. Any male or female patient aged 18 or older
2. Able to provide serum and urine specimen before treatment
3. Diagnosis with benign disease of the urinary system, such as urinary calculi and benign prostatic hyperplasia.

Exclusion Criteria:

1. Kidney and liver dysfunction.
2. Incomplete clinical information and laboratory test result
3. Tumor-related treatment was received preoperatively
4. Preoperative routine examination and medical history indicate a history of diabetes, hyperlipidemia and other metabolic diseases or other malignant tumors

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bladder cancer or benign. disease of urinary system will be enrolled.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 1 year
  Measurement the sensitivity of diagnostic model based on urine and serum metabolomics in differentiating between bladder cancer and benign disease of the urinary system
Specificity | 1 year
  Measurement the specificity of diagnostic model based on urine and serum metabolomics in differentiating between bladder cancer and benign disease of the urinary system

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University